CLINICAL TRIAL: NCT01414595
Title: Molecular Characterization of Lung Cancer: A Collaboration With the Cancer Genome Atlas Project (TGCA)
Brief Title: Study of Tissue Samples From Patients With Non-Small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-151107; CALGB-151107; CDR0000706375 (Registry Identifier: NCI Physician Reference Desk)
Record Dates: First submitted 2011-08-10; First posted 2011-08-11 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Lung Cancer
Keywords: adenocarcinoma of the lung; adenosquamous cell lung cancer; non-small cell lung cancer; squamous cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung | interventions — DNA Methylation; Gene Expression Profiling; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tumor and blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: CALGB 140202 outlines the standard procedures for sample procurement. Samples to be used for this project have already been obtained and are currently banked at the CALGB Pathology Coordinating Office (PCO) and the Lung Cancer Tissue Bank at Brigham and Women's Hospital.
  Interventions: Genetic: DNA analysis; Genetic: DNA methylation analysis; Genetic: RNA analysis; Genetic: gene expression analysis; Genetic: polymorphism analysis; Other: laboratory biomarker analysis; Other: medical chart review

INTERVENTIONS:
Genetic: DNA analysis
Genetic: DNA methylation analysis
Genetic: RNA analysis
Genetic: gene expression analysis
Genetic: polymorphism analysis
Other: laboratory biomarker analysis
Other: medical chart review

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research trial studies tissue samples from patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To identify and characterize single nucleotide variations (SNVs) in non-small cell lung cancer (NSCLC) specimens.
* To identify and characterize structural variations in the genomes of NSCLC specimens.
* To identify and characterize other genomic alterations including, but not limited to, expression profiling and methylation.

OUTLINE: DNA and RNA extracted from archived specimens are analyzed for single nucleotide variations, structural variations in the genomes, and other genomic alterations including, but not limited to, gene expression profiling and methylation. Clinical data related to disease, treatment, and recurrence from each patient sample is also collected.

ELIGIBILITY:
* Patient must have been registered to CALGB 140202.
* Tumor histology should be either primary adenocarcinoma or squamous cell carcinoma of the lung.
* Patients are eligible for this study if their samples from CALGB 140202 are available.
* All living patients must sign the CALGB 151107 consent form to be eligible for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with lung cancer who are registered to CALGB-140202.
Sampling Method: Non-Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2012-03; Primary Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Identification and characterization of SNVs in primary adenocarcinoma of the lung or squamous cell carcinoma of the lung | up to 5 years
Identification and characterization of structural variations in the genomes of NSCLC | up to 5 years
Identification and characterization of other genomic alterations including, but not limited to, gene expression profiling and methylation | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ramaswamy Govindan, MD, Study Chair — Washington University School of Medicine
Locations (11):
- United States (11):
  - Samuel Oschin Comprehensive Cancer Institute at Cedars-Sinai Medical Center, Los Angeles, California
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Duke Cancer Institute, Durham, North Carolina
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island